CLINICAL TRIAL: NCT03200418
Title: Evaluation of the Effect of Output on Newly Developed Adhesives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_10_11
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Ileostomy - Stoma
MeSH Terms: interventions — Cyclin-Dependent Kinase Inhibitor p15; Cyclin-Dependent Kinase Inhibitor p16

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of new adhesives (Experimental): On the peristomal area four different patches are applied to the skin. There is a bag welded on each patch. The bag contains real output.
  The difference between the four patches is that they consist of different adhesives.
  One patch is made of a standard hydrocolloid adhesive
  The primary endpoint is maesured after 8 hours and 24 hours And the three other patches consist of the newly developed adhesives. P-4 P-15 P-16
  Interventions: Other: Standard hydrocolloid adhesive; Other: P-4; Other: P-15; Other: P-16

INTERVENTIONS:
Other: Standard hydrocolloid adhesive — This patch is made of standard hydrocolloid adhesive
Other: P-4 — This patch is made of new adhesive
Other: P-15 — This patch is made of new adhesive
Other: P-16 — This patch is made of new adhesive

SUMMARY:
The study investigates the impact real output has on the adhesion of the adhesives.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had a stoma for more than one year
4. Have intact skin on the area used in the evaluation
5. Has a stoma with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tab-let/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Actively participating in other interventional clinical investigations or have previously participated in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 8 hours
  The trans epidermal water loss is measured on the peristomal skin using a probe. The trans epidermal water loss is a measure for the skins barrier function. There is always a loss of water from the skin due to natural evaporation. However, when the skin barrier is damaged the evaporation of water increases leading to a higher trans epidermal water loss. Thus, trans epidermal water loss is used to assess the damage to the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No